CLINICAL TRIAL: NCT01518075
Title: Breathing-swallowing Interaction in Chronic Obstructive Pulmonary Disease (COPD) Patients Hospitalized in Intensive Care Unit for an Acute Exacerbation: Impact of Non Invasive Ventilation. Physiological Evaluation
Brief Title: Breathing-swallowing Interaction in Chronic Obstructive Pulmonary Disease Patients - Impact of Non Invasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DEGLUT
Record Dates: First submitted 2012-01-21; First posted 2012-01-25 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Decompensated COPD With (Acute) Exacerbation
Keywords: Chronic Obstructive Pulmonary Disease; Non invasive mechanical ventilation; Breathing-swallowing interaction; Intensive Care Unit
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non invasive mechanical ventilation (Experimental): Evaluation of breathing swallowing interaction under non invasive mechanical ventilation
  Interventions: Other: Non Invasive Mechanical Ventilation
- Spontaneous Breathing (Active Comparator): Evaluation of breathing swallowing interaction without non invasive mechanical ventilation
  Interventions: Other: Spontaneous Breathing

INTERVENTIONS:
Other: Spontaneous Breathing — Evaluation of breathing - swallowing interaction without non invasive mechanical ventilation. Patient breath spontaneously.
  Measurements of respiratory and swallowing parameters were monitored using respiratory inductive plethysmography. Swallowing was monitored noninvasively. Two bolus sizes were used, (5, 10 ml), in random order. Five sets of two boluses were studied, taking care not to use the same bolus size twice consecutively. The study participants were blinded to bolus size.
  Other Names: SB
  Arms: Spontaneous Breathing
Other: Non Invasive Mechanical Ventilation — Evaluation of breathing - swallowing interaction with non invasive mechanical ventilation. Patient breath under non invasive mechanical ventilation. Measurements of respiratory and swallowing parameters were monitored using respiratory inductive plethysmography. Swallowing was monitored noninvasively. Two bolus sizes were used, (5, 10 ml), in random order. Five sets of two boluses were studied, taking care not to use the same bolus size twice consecutively. The study participants were blinded to bolus size.
  Other Names: NIV
  Arms: Non invasive mechanical ventilation

SUMMARY:
In the investigators' knowledge there are no data about the impact of non invasive mechanical ventilation on the breathing-swallowing interaction.

Our main objective is to evaluate breathing-swallowing interaction in Chronic Obstructive Pulmonary Disease (COPD) patients hospitalized in intensive care unit for an acute exacerbation, and evaluate the impact of using non invasive mechanical ventilation (NIV)

DETAILED DESCRIPTION:
In healthy subjects previous studies showed that most swallows started during expiration and were followed by expiration, a pattern believed to contribute to airway protection during swallowing. However In healthy individuals, the occurrence of inspiration after swallows was increased by hypercapnia or application of an inspiratory elastic load.

In a previous study the investigators have demonstrated that patients with neuromuscular disorders exhibited piecemeal deglutition leading to an increase in the time needed to swallow a water bolus, as well as occurrence of inspiration after nearly half the swallows. These abnormalities which increased with the decreasing of respiratory muscle performances may explain feeding difficulties. However in tracheostomized patients who could breathe spontaneously, piecemeal deglutition and swallowing time per bolus were diminished by the use of mechanical ventilation.

In the investigators' knowledge there are no data about the impact of non invasive mechanical ventilation on the breathing-swallowing interaction.

The investigators' main objective is to evaluate breathing-swallowing interaction in Chronic Obstructive Pulmonary Disease (COPD) patients hospitalized in intensive care unit for an acute exacerbation, and evaluate the impact of using non invasive mechanical ventilation (NIV)

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Obstructive Pulmonary Disease
* Age > 18 years
* Hospitalized in Intensive care for an acute exacerbation
* Requiring Non invasive mechanical ventilation
* Able to breath spontaneously without non invasive ventilation more than 4h/day
* Without bulbar dysfunction

Exclusion Criteria:

* Hemodynamic instability
* Absence of consent
* Severe Hypoxemia
* pH < 7,30
* No cooperation of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Impact of non invasive mechanical ventilation on breathing swallowing interaction | 2 h
  Physiological evaluation of breathing - swallowing interaction with or without non invasive mechanical ventilation

SECONDARY OUTCOMES:
Correlation between breathing swallowing interaction and functional respiratory parameters | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas TERZI, MD - PhD, Principal Investigator — University Hospital, Caen; Frédéric Lofaso, MD-PhD, Principal Investigator — University Hospital, Garches
Locations (1):
- University Hospital, Caen, Caen, France